CLINICAL TRIAL: NCT00000851
Title: Trial of Stavudine (d4T) Plus Didanosine (ddI) in Children on Long-Term Stavudine Monotherapy, and Stavudine Versus Stavudine Plus Didanosine in Children on Long-Term Zidovudine Monotherapy: A Rollover Protocol for ACTG 240 Participants and Children Receiving Prescription Zidovudine
Brief Title: Comparison of Stavudine Used Alone or in Combination With Didanosine in HIV-Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 327; 11300 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Antiviral Agents; Stavudine
MeSH Terms: conditions — HIV Infections | interventions — Stavudine; Didanosine

INTERVENTIONS:
Drug: Stavudine
Drug: Didanosine

SUMMARY:
To evaluate the safety and determine the pharmacokinetic disposition of stavudine (d4T) alone and in combination with didanosine (ddI), and whether concurrent administration alters the disposition of either drug. To compare d4T versus d4T plus ddI with respect to short and long term changes from baseline in plasma HIV RNA concentrations. To determine the relationship, if any, between drug exposure and viral burden.

In a pilot study of d4T and ddI given to eight children with advanced HIV for 24 weeks, the three children with baseline counts greater than 50 cells/micro liter experienced a 20% increase in their CD4+ lymphocyte counts. Based on these results, controlled trials of the same regimen for children with less advanced HIV disease should be undertaken.

DETAILED DESCRIPTION:
In a pilot study of d4T and ddI given to eight children with advanced HIV for 24 weeks, the three children with baseline counts greater than 50 cells/micro liter experienced a 20% increase in their CD4+ lymphocyte counts. Based on these results, controlled trials of the same regimen for children with less advanced HIV disease should be undertaken.

Eligible subjects receiving d4T will be assigned in an open manner to Arm 1, and subjects who have been receiving zidovudine (AZT) will be assigned in a randomized, double blind manner to Arms 2 and 3. Each subject will receive study drug for 48 weeks as follows: Arm 1 - d4T plus ddI, Arm 2 - d4T alone, Arm 3 - d4T plus ddI.

ELIGIBILITY:
Inclusion Criteria

Patients must:

* Be on-study, on-treatment in ACTG 240, or receiving AZT monotherapy by prescription for at least 6 months immediately preceding enrollment.
* Have laboratory evidence of HIV-1 infection < 18 months - 2 positive viral tests >= 18 months - 2 positive viral tests or 2 or more positive tests for HIV antibody
* Have parent or legal guardian willing to sign a consent.

Prior Medication: Required:

* On-study, on-treatment in ACTG 240 (D4T or AZT) or receiving AZT monotherapy by prescription for at least six months immediately preceding this trial.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Intractable diarrhea or vomiting.
* Current clinical or laboratory Grade 3 or worse toxicities.

Concurrent Medication:

Excluded:

* Concurrent use of antiretroviral agents other than those provided by the study, immunomodulators (other than IVIG or corticosteroids), or other investigational drugs except for those in ACTG 254 and ACTG 219.
* Chemotherapy for active malignancy.

Patients with any of the following prior conditions are excluded:

* Reached an ACTG 240 defined endpoint, or are permanently off ACTG 240 study treatment.
* Prescription AZT recipients may not have received > 6 weeks of d4T or ddI previously.
* Subjects who have had chemotherapy for active malignancy.

Prior Medication:

Excluded:

* Prescription AZT recipients may not have received > 6 weeks of d4T or ddI previously.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kline M, Study Chair; Van Dyke R, Study Chair
Locations (35):
- United States (32):
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Univ. of Connecticut Health Ctr., Dept. of Ped., Farmington, Connecticut
  - Connecticut Children's Med. Ctr., Hartford, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Cook County Hosp., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - Children's Med. Ctr. Dallas, Dallas, Texas
  - Texas Children's Hosp. CRS, Houston, Texas
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Kline MW, Van Dyke RB, Lindsey JC, Gwynne M, Culnane M, Diaz C, Yogev R, McKinney RE Jr, Abrams EJ, Mofenson LM. Combination therapy with stavudine (d4T) plus didanosine (ddI) in children with human immunodeficiency virus infection. The Pediatric AIDS Clinical Trials Group 327 Team. Pediatrics. 1999 May;103(5):e62. doi: 10.1542/peds.103.5.e62. PMID 10224206
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891